CLINICAL TRIAL: NCT05818189
Title: Cortical Correlates of Gait in Parkinson's Disease: Impact of Medication and Cueing
Acronym: cueing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Martina Mancini, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01HD110389 (NIH); R01HD110389 (NIH)
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
Keywords: Tactile cueing; Gait; Turning; Cortical activity
MeSH Terms: conditions — Parkinson Disease | interventions — Precision Medicine

STUDY DESIGN:
Intervention Model Description: 60 participants with PD from Aim I, will be randomized into one, of two, cueing interventions: 1) personalized, step-synchronized tactile cueing and 2) tactile cueing at fixed intervals as an active control group. We will analyze the immediate effects of the cueing intervention on gait automaticity. In addition, we will explore the feasibility and potential benefits of independent use of tactile cueing during a week in daily life for a future clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The subjects will not know which intervention is favored for improving gait automaticity and the researchers analyzing the data will not know which intervention group subjects were randomly assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized cueing (Experimental): Personalized, step-synchronized tactile cueing, enhancing proprioceptive inputs, in the form of real-time, closed-loop tactile feedback signaling left and right stance times while walking
  Interventions: Device: Personalized tactile cueing
- Fixed cueing (Active Comparator): Tactile cueing at fixed intervals, enhancing proprioceptive inputs, in the form of open-loop tactile feedback (fixed rhythm) signaling left and right stance times while walking
  Interventions: Device: Fixed tactile cueing

INTERVENTIONS:
Device: Personalized tactile cueing — We will use as an external cue, a system of tactile cueing with the purpose of enhancing proprioceptive inputs, in the form of real-time(synchronized to the gait heel strike), closed-loop tactile feedback signaling left and right stance times while walking. Also, the participants use the same system cueing in closed-loop feedback during daily life for one week.
  Other Names: personalized
  Arms: Personalized cueing
Device: Fixed tactile cueing — We will use as an external cue, a system of tactile cueing with the purpose of enhancing proprioceptive inputs, in the form of real-time, open-loop(fixed rhythm) tactile feedback signaling left and right stance times while walking. Also, the participants use the same system cueing in open-loop feedback during daily life for one week.
  Other Names: fixed
  Arms: Fixed cueing

SUMMARY:
The purpose of the study is to determine the effects of a novel, personalized, tactile cueing system on gait automaticity. The researchers hypothesized that step-synchronized tactile cueing will reduce prefrontal cortex activity (improve automaticity) and improve gait variability (as well as gait speed). The researchers predict that improved automaticity with improved gait variability will be associated with increased activation of other than prefrontal cortical areas while walking (i.e., sensory-motor). To determine the effects of cueing, 60 participants with PD from will be randomized into one, of two, cueing interventions: 1) personalized, step-synchronized tactile cueing and 2) tactile cueing at fixed intervals as an active control group. In addition, the researchers will explore the feasibility and potential benefits of independent use of tactile cueing during a week in daily life for a future clinical trial.

This project will characterize the cortical correlates of gait automaticity, the changes in gait automaticity with cueing in people with Parkinson's Disease, and how these changes translate to improvement in gait and turning. The long-term goal is to unravel the mechanisms of impaired gait automaticity in Parkinson's Disease.

DETAILED DESCRIPTION:
Cortical correlates of gait automaticity in Parkinson's disease: impact of cueing

A well-recognized hallmark of healthy walking is automaticity, defined as the ability of the nervous system to successfully coordinate movement with minimal use of attention-demanding, executive resources. It has been proposed that many walking abnormalities in people with Parkinson's disease (PD) are characterized by a shift in locomotor control from healthy automaticity to compensatory, executive control. This shift to less automaticity is potentially detrimental to walking performance as executive control strategies are not optimized for locomotor control, place excessive demands on a limited cognitive reserve, and continuously require attention. It has been hypothesized that as gait becomes more variable, as in people with Parkinson's Disease, control of gait is less automatic, i.e., requires more prefrontal cortex involvement. However, as gait variability is not a direct measure of automaticity, it is controversial whether it truly reflects impaired gait automaticity or impaired gait stability (i.e., dynamic balance). The recent development of wireless, functional, near-infrared spectroscopy (fNIRS) of the brain provides more direct, physiological measures of automaticity, such as reduced prefrontal cortex activity. However, the contribution of other cortical areas to the concept of gait automaticity is largely unknown. Here, for the first time, the researchers will use a full cap fNIRS system to monitor cortical activity in multiple brain areas and wearable, inertial sensors to determine how cognitive abilities, levodopa, and cueing influence gait automaticity.

The effects of cognitive dysfunction and interventions on gait in people with Parkinson's Disease are complex. Impaired executive function has been associated with impaired gait and balance in PD, but it is not known if this relationship is due to the inability to compensate for poor basal ganglia control of gait automaticity with increased prefrontal cortex activity while walking. Sensory cueing may increase gait speed and reduce prefrontal activity but unlike levodopa, it may result in reduced gait variability due to enhanced automaticity. The researchers recently developed a novel type of personalized (triggered by the subject's own walking pattern), step-synchronized tactile stimulation on the wrists to improve the quality of gait and turning in people with Parkinson's Disease. The researchers will now compare the effects of cognitive dysfunction, dopaminergic medication, and tactile cueing on the quality of gait and turning and investigate whether improvements reflect changes in prefrontal activity.

This project will characterize the cortical correlates of gait automaticity, the changes in gait automaticity with cueing in people with PD, and how these changes translate to improvement in gait and turning. The long-term goal is to unravel the mechanisms of impaired gait automaticity in Parkinson's Disease.

The purpose of the study is to determine the effects of a novel, personalized, tactile cueing system on gait automaticity. The researchers hypothesized that step-synchronized tactile cueing will reduce prefrontal cortex activity (improve automaticity) and improve gait variability (as well as gait speed). We predict that improved automaticity with improved gait variability will be associated with increased activation of other than prefrontal cortical areas while walking (i.e., sensory-motor). To determine the effects of cueing, 60 participants with PD from will be randomized into one, of two, cueing interventions: 1) personalized, step-synchronized tactile cueing and 2) tactile cueing at fixed intervals as an active control group. A secondary analysis will explore whether the effect of cueing on gait automaticity is influenced by cognitive dysfunction. In addition, we will explore the feasibility and potential benefits of independent use of tactile cueing during a week in daily life for a future clinical trial. We will explore feasibility and efficacy of cueing in daily life comparing data of gait and turning from a week of continuous monitoring without and with using the tactile cueing. In addition, we will test whether any retention on gait and turning is present by adding a third week of continuous monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's Disease from movement disorders neurologist with the United Kingdom Brain Bank criteria of bradykinesia with 1 or more of the following - rest tremor, rigidity, and balance problems not from visual, vestibular, cerebellar or proprioceptive conditions
* Without musculoskeletal or peripheral or central nervous system disorders (other than PD) that could significantly affect their balance and gait
* All subjects will be capable of following directions for the protocols and to give informed consent.
* Hoehn & Yahr Levels II-III.

Exclusion Criteria:

* Severe dyskinesia that may affect quality of fNIRS.
* Major musculoskeletal or neurological disorders, structural brain disease, epilepsy, acute illness or health history, other than Parkinson's Disease, significantly affecting gait and turning i.e., peripheral neuropathy with proprioceptive deficits (detected as lack of toe proprioception assessed during the neurological exam at Day 1), musculoskeletal disorders, vestibular problem, head injury, stroke.
* Montreal cognitive assessment (MoCA) score < 21 or dementia that precludes consent to participate or ability to follow testing procedures
* Inability to stand or walk for 2 minutes without an assistive device.
* Idiopathic Parkinson's Disease exclusion criteria: Parkinson plus syndromes such as progressive supranuclear palsy, multiple system atrophy, or corticobasal syndrome or implanted electrodes for deep brain stimulation (DBS), possible vascular parkinsonism, current use of dopamine-blocking agents or cholinesterase inhibitor (as may affect Prefrontal cortical activity while walking).

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Prefrontal cortex activity | day 1
  Oxygenated hemoglobin over the prefrontal cortex measures by fNIRS
Parietal cortex activity | day 1
  Oxygenated hemoglobin over the parietal cortex measures by fNIRS
Stride time variability | day 1
  Variability of stride time during 2 minute walking
Local Dynamic Stability | day 1
  Stability during gait is assessed by phase dependent local dynamic stability (LDS) measures of the trunk acceleration while walking
Turn duration | day 1
  Average duration of 360 turning while performing a 1 minute turning in place task
Turn jerk | day 1
  Average turning smoothness while performing a 1 minute turning in place task

SECONDARY OUTCOMES:
Supplementary motor area cortical activity | day 1
  Oxygenated hemoglobin over the SMA cortex measures by fNIRS
Occipital cortical activity | day 1
  Oxygenated hemoglobin over the visual cortex measures by fNIRS
Gait speed | day 1
  Average gait speed during 2 minute walking
Gait speed variability | day 1
  Variability of gait speed during 2 minute walking
Stride time | day 1
  Average stride duration during 2 minute walking
Stride length | day 1
  Average stride length during 2 minute walking
Stride length variability | day 1
  Variability of stride length during 2 minute walking
Turn duration variability | day 1
  Variability of turning duration while performing a 1 minute turning in place task
Turn jerk variability | day 1
  Variability of turning smoothness while performing a 1 minute turning in place task
Number of steps during turning | day 1
  Average number of steps while performing a 1 minute turning in place task
Number of steps during turning variability | day 1
  Variability of number of steps while performing a 1 minute turning in place task
Turn velocity | day 1
  Average turning velocity while performing a 1 minute turning in place task
Turn velocity variability | day 1
  Variability of turning velocity while performing a 1 minute turning in place task

CONTACTS AND LOCATIONS:
Overall Officials: Martina Mancini, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, we can share de-identified data related to study outcomes measures.
Supporting Information: Study Protocol, SAP
Time Frame: Data would be available 6 months after the end of data collection. Data will be stored in our laboratory data repository and so will be available indefinitely.
Access Criteria: Data will not be stored on a public website, however researchers may contact us for access to the data. We will send data electronically via a secure server.

REFERENCES:
- [Derived] Burgos PI, Liu W, Silva-Batista C, Baker-Alcala F, Carlson-Kuhta P, King LA, Horak FB, Chung KA, Lapidus JA, Mancini M. Personalized versus fixed tactile cueing in Parkinson's disease: Protocol for a randomized controlled trial on gait automaticity. PLoS One. 2025 Nov 21;20(11):e0336859. doi: 10.1371/journal.pone.0336859. eCollection 2025. PMID 41270079